CLINICAL TRIAL: NCT03239171
Title: Combination of Cancer Ablation and Life Information Rehabilitation Therapy for Unresectable Lung Cancer
Brief Title: Bioinformation Therapy for Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shengxin Biotechnology Institute, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bioinformation-lung
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2017-08

CONDITIONS: Small-cell Lung Cancer
Keywords: Cancer ablation; Life information rehabilitation therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cryosurgery; Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cancer ablation (Active Comparator): In this group, the patients will receive ablation therapy (e.g. cryosurgery or irreversible electroporation) first for big tumors (> 2 cm). The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Cancer ablation
- Life information rehabilitation therapy (Active Comparator): In this group, the patients will drink "Qilisheng" Immunoregulatory Oral Solution for consecutive 3 months. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Life information rehabilitation therapy
- Combination therapy (Experimental): In this group, the patients will receive the combination therapy including ablation and life information rehabilitation therapy. The ablation therapy (e.g. cryosurgery or irreversible electroporation) will be performed first for big tumors (> 2 cm), then "Qilisheng" Immunoregulatory Oral Solution will be provided for consecutive 3 months. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Cancer ablation; Drug: Life information rehabilitation therapy
- Control (No Intervention): In this group, the patients will receive no special treatment and as a control group. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).

INTERVENTIONS:
Device: Cancer ablation — Tumors bigger than 2 cm are fit for ablation therapy, percutaneously under CT scan or ultrasound.
  Other Names: Cryoablation or irreversible electroporation
  Arms: Cancer ablation; Combination therapy
Drug: Life information rehabilitation therapy — Each treatment: one bottle solution each day, consecutive 3 months, oral administration
  Other Names: "Qilisheng" Immunoregulatory Oral Solution
  Arms: Combination therapy; Life information rehabilitation therapy

SUMMARY:
The aim of this study is the synergistic effect of cancer ablation and life information rehabilitation therapy on unresectable lung cancer.

DETAILED DESCRIPTION:
By enrolling patients with unresectable lung cancer adapted to enrolled criteria, this study will document for the first time the synergistic effect of cancer ablation and life information rehabilitation therapy. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies
* Body tumor 1-6, with at least one tumor length > 2 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Relief degree of tumors | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
  The duration between treatment and cancer recurrence
Overall survival（OS） | 3 years
  The duration between treatment and patient pass away

CONTACTS AND LOCATIONS:
Locations (1):
- Fuda cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China